CLINICAL TRIAL: NCT00871728
Title: Change in SCIO (Scoring Clinical Index For Onychomycosis) in Toenail Onychomycosis Treating With Itraconazole Capsules
Brief Title: Scoring Clinical Index For Onychomycosis in Toenail Onychomycosis Treating With Itraconazole Capsules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013837; ITR-KOR-4078
Record Dates: First submitted 2009-02-13; First posted 2009-03-30 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Onychomycosis, Toe
Keywords: Onychomycosis, Toe; Itraconazole; Sporanox
MeSH Terms: conditions — Onychomycosis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Itraconazole (Experimental)
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Itraconazole (ICZ) capsule will be administered in 3 cycles (Week 1, Week 5 and Week 9) and each cycle will consist of taking 2 capsules of 100 milligram (mg) each, orally twice daily, continuously for 1 week and then not taking medication for next 3 weeks. Total duration of treatment will be 49 weeks.
  Other Names: Sporanox

SUMMARY:
The purpose of this study is to evaluate the participants with toenail onychomycosis (fungal infection of the nail) confirmed positive by potassium hydroxide (KOH) and bacterial identification test after administration of itraconazole (ICZ) capsule, to identify the change in Scoring Clinical Index for Onychomycosis (SCIO) score and to determine the relationship between the change of SCIO score and mycological cure rate and clinical improvement.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (when more than one hospital or medical school team work on a medical research study) study of ICZ in participants with onychomycosis. The present study consists of 2 periods: Screening period (up to Week minus 2) and Treatment period (up to Week 49). The ICZ will be administered in 3 cycles (Week 1, Week 5 and Week 9) and each cycle will consist of taking 2 capsules of 100 milligram (mg) each, orally, twice daily, continuously for 1 week. Total duration of treatment will be of 49 weeks. Efficacy will primarily be evaluated by percentage of participants showing 10 percent or higher response in SCIO Score. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Onychomycosis participants whose etiologic agent is identified by potassium hydroxide (KOH) smear and bacterial identification test
* Participants with Scoring Clinical Index for Onychomycosis (SCIO) greater than or equal to 9
* Participants who are healthy in general in following items: medical and medication history, physical examination before administration time, vital signs (blood pressure and pulse) and clinical laboratory tests (clinical test results [liver function and renal function] are within 2 times the normal range)
* Female participants of child-bearing age who use acceptable contraceptives
* Participants who can understand features of clinical study and signed informed consent form

Exclusion Criteria:

* Participants with psoriasis (scaly skin rash)
* Diabetic participants who take an anti-diabetic drug
* Pregnant or breast feeding female participants
* Participants with clinical evidence of arterial insufficiency or peripheral vascular disease and medical history of decreased ventricular function like congestive heart failure (heterogeneous condition in which the heart is unable to pump out sufficient blood to meet the metabolic need of the body)
* Participants who applied a topical antifungal agent (nail lacquer) on target nail within 1 month before the study medication administration and who took an oral antifungal agent within 3 month before the study medication administration

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole: Itraconazole (ICZ) capsule was administered in 3 cycles (Week 1, Week 5 and Week 9) and each cycle consists of taking 2 capsules of 100 milligram (mg) each, orally twice daily, continuously for 1 week and then not taking medication for next 3 weeks. Total duration of treatment was 49 weeks.
Period: Overall Study
Arm/Group | Itraconazole
Started | 132
Treated | 130
Completed | 112
Not Completed | 20
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 7
Not completed — Lost to Follow-up | 2
Not completed — Failed to Visit Hospital | 4
Not completed — Participant Non-compliance | 1
Not completed — Withdrawal of Informed Consent | 5

BASELINE CHARACTERISTICS:
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
Age Continuous [Mean (Standard Deviation); unit: years] — Data presented only for 117 participants as they were part of Full Analysis Set (FAS) population.
  years | 44.6 (10.42)
Sex: Female, Male [Count of Participants; unit: Participants] — Data presented only for 117 participants as they were part of FAS population.
  Participants
    Female | 47
    Male | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Showing 10 Percent or Higher Response in Scoring Clinical Index for Onychomycosis (SCIO) Score at Week 5
Description: The SCIO is based on clinical state and its items include major factors that can have an effect on the outcome of onychomycosis treatment. The factors include the clinical form, depth of an infected area and subungal hyperkeratosis. The SCIO score range from 1 to 30 and higher score indicates more severity. The score is classified into 7 steps and as there is treatment for each step, treatment based on the clinical state can be applied consistently. Percentage of participants who show an improvement in SCIO score by 10 percent or more at Week 5 compared to Baseline were reported.
Time Frame: Baseline and Week 5
Population: The Full analysis set (FAS) population included all participants except for those participants who violated the major selection and exclusion criteria or did not take the study medication even once or those participants who didn't participate in Week 5 assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
percentage of participants | 25.6

2. Primary Outcome: Percentage of Participants Showing 10 Percent or Higher Response in Scoring Clinical Index for Onychomycosis (SCIO) Score at Week 9
Description: The SCIO is based on clinical state and its items include major factors that can have an effect on the outcome of onychomycosis treatment. The factors include the clinical form, depth of an infected area and subungal hyperkeratosis. The SCIO score range from 1 to 30 and higher score indicates more severity. The score is classified into 7 steps and as there is treatment for each step, treatment based on the clinical state can be applied consistently. Percentage of participants who show an improvement in SCIO score by 10 percent or more at Week 9 compared to Baseline were reported.
Time Frame: Baseline and Week 9
Population: The FAS population included all participants except for those participants who violated the major selection and exclusion criteria or did not take the study medication even once or those participants who didn't participate in Week 5 assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
percentage of participants | 50.4

3. Primary Outcome: Percentage of Participants Showing 10 Percent or Higher Response in Scoring Clinical Index for Onychomycosis (SCIO) Score at Week 13
Description: The SCIO is based on clinical state and its items include major factors that can have an effect on the outcome of onychomycosis treatment. The factors include the clinical form, depth of an infected area and subungal hyperkeratosis. The SCIO score range from 1 to 30 and higher score indicates more severity. The score is classified into 7 steps and as there is treatment for each step, treatment based on the clinical state can be applied consistently. Percentage of participants who show an improvement in SCIO score by 10 percent or more at Week 13 compared to Baseline were reported.
Time Frame: Baseline and Week 13
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
percentage of participants | 80.3

4. Primary Outcome: Percentage of Participants Showing 10 Percent or Higher Response in Scoring Clinical Index for Onychomycosis (SCIO) Score at Week 25
Description: The SCIO is based on clinical state and its items include major factors that can have an effect on the outcome of onychomycosis treatment. The factors include the clinical form, depth of an infected area and subungal hyperkeratosis. The SCIO score range from 1 to 30 and higher score indicates more severity. The score is classified into 7 steps and as there is treatment for each step, treatment based on the clinical state can be applied consistently. Percentage of participants who show an improvement in SCIO score by 10 percent or more at Week 25 compared to Baseline were reported.
Time Frame: Baseline and Week 25
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
percentage of participants | 84.6

5. Primary Outcome: Percentage of Participants Showing 10 Percent or Higher Response in Scoring Clinical Index for Onychomycosis (SCIO) Score at Week 37
Description: The SCIO is based on clinical state and its items include major factors that can have an effect on the outcome of onychomycosis treatment. The factors include the clinical form, depth of an infected area and subungal hyperkeratosis. The SCIO score range from 1 to 30 and higher score indicates more severity. The score is classified into 7 steps and as there is treatment for each step, treatment based on the clinical state can be applied consistently. Percentage of participants who show an improvement in SCIO score by 10 percent or more at Week 37 compared to Baseline were reported.
Time Frame: Baseline and Week 37
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
percentage of participants | 86.3

6. Primary Outcome: Percentage of Participants Showing 10 Percent or Higher Response in Scoring Clinical Index for Onychomycosis (SCIO) Score at Week 49
Description: The SCIO is based on clinical state and its items include major factors that can have an effect on the outcome of onychomycosis treatment. The factors include the clinical form, depth of an infected area and subungal hyperkeratosis. The SCIO score range from 1 to 30 and higher score indicates more severity. The score is classified into 7 steps and as there is treatment for each step, treatment based on the clinical state can be applied consistently. Percentage of participants who show an improvement in SCIO score by 10 percent or more at Week 49 compared to Baseline were reported.
Time Frame: Baseline and Week 49
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
percentage of participants | 80.3

7. Secondary Outcome: Percentage of Participants Showing Mycological Cure
Description: Mycological cure was defined as a case in which the results of both potassium hydroxide (KOH) smear test and bacterial identification test (BIT) were found to be negative at each pre-defined time point.
Time Frame: Week 13, 25, 37 and 49
Population: The FAS population, missing values imputed using last observation carried forward (LOCF) method. 'n' included those participants who were evaluable for this measure at specific time points.
Measure: Number; unit: percentage of participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 117
percentage of participants
  Negative KOH Smear Test : Week 13 (n=109) | 70.6
  Negative KOH Smear Test : Week 25 (n=103) | 83.5
  Negative KOH Smear Test : Week 37 (n=102) | 90.2
  Negative KOH Smear Test : Week 49 (n=99) | 83.8
  Negative BIT : Week 13 (n=108) | 64.8
  Negative BIT : Week 25 (n=103) | 79.6
  Negative BIT : Week 37 (n=102) | 81.4
  Negative BIT : Week 49 (n=97) | 82.5

ADVERSE EVENTS:
Time Frame: From Screening up to 49 weeks
Arm/Group | Itraconazole
Serious Adverse Events (participants affected / at risk) | 1/130
Other Adverse Events (participants affected / at risk) | 35/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole (N=130)
Dyspepsia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole (N=130)
Dyspepsia (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Acute tonsillitis (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sputum (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Adverse event (General disorders) | 3
Oedema peripheral (General disorders) | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Pyuria (Renal and urinary disorders) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Mucopolysaccharidosis (Congenital, familial and genetic disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1

LIMITATIONS AND CAVEATS:
Initially it was planned to assess clinical cure rate but analysis for clinical cure rate following the administration of the study drug was replaced by change in SCIO scores which was the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot provide any trial related information to external parties' without mutual agreement with the sponsor. This is valid even after the contract is canceled.